CLINICAL TRIAL: NCT01974791
Title: GET Living: Graded Exposure Treatment for Children and Adolescents With Chronic Pain
Acronym: GET Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Laura Simons(Giardi), Staff Psychologist, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00007276; 82267 (Other Grant/Funding Number: American Pain Society)
Record Dates: First submitted 2013-10-22; First posted 2013-11-04 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Chronic Pain; Neuralgia; Musculoskeletal Pain; Headache
MeSH Terms: conditions — Chronic Pain; Neuralgia; Musculoskeletal Pain; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GET Living Treatment (Experimental)
  Interventions: Behavioral: GET Living

INTERVENTIONS:
Behavioral: GET Living — GET Living is an exposure based treatment jointly delivered by a cognitive-behavioral therapist and physical therapy to help children and adolescents suffering with chronic pain and headache progressively return to valued life activities.

SUMMARY:
The broad aim of the study is to implement and evaluate the efficacy of Graded Exposure Treatment (GET Living) to target elevated pain-related fears in children with chronic pain. Pain-related fear is an important psychological factor associated with poor outcomes in children suffering with chronic pain. To examine the efficacy of GET Living in addressing pain-related fears the investigators propose to use a sequential replicated randomized single-case experimental phase design with multiple measures. The specific aims are to 1) evaluate the effectiveness and acceptability of individually tailored GET Living for children with high pain-related fear and functional disability and 2) define anatomical and resting state connectivity patterns in the brains of children and adolescents with complex chronic pain prior to and after participation in GET Living.

ELIGIBILITY:
Inclusion Criteria:

* Pain-related fear (score >40 on the Fear of Pain Questionnaire (FOPQ (Simons et al., 2011a))
* Musculoskeletal, neuropathic limb or back pain, or headache
* Functional limitations (score > 12 on the Functional Disability Inventory (FDI (Kashikar-Zuck et al., 2001; Walker and Greene, 1991)).

Exclusion Criteria:

* Significant cognitive impairment (e.g., intellectual disability)
* Serious psychopathology (e.g., active suicidality).
* Acute trauma (e.g., spondylolithesis, disk herniation, fracture, acute tendonitis)
* Systemic disease in active inflammatory state
* Biomechanical deficit that would limit ability to engage in exposure activities (e.g. severe muscle atrophy)
* Making gains in current physical therapy or have not had physical therapy, but it is clearly indicated

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2013-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Decrease in Fear of Pain | Decrease in Fear of Pain from Baseline to end of treatment at 6-weeks, on average

SECONDARY OUTCOMES:
Decrease in Functional Disability | Decrease in Functional Disability from Baseline to end of treatment at 6-weeks, on average
Improvement in School Functioning | Improvement in School Functioning from baseline to end of treatment at 6-weeks, on average
Decrease in Pain Catastrophizing | Decrease in Pain Catastrophizing from baseline to end of treatment at 6-weeks, on average
Decrease in Pain Intensity | Decrease in Pain Intensity from baseline to end of treatment at 6-weeks, on average
Increase in Physical Activity | Increase in Physical Activity from baseline to end of treatment at 6-weeks, on average

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Simons, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital Waltham, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Schemer L, Hess CW, Van Orden AR, Birnie KA, Harrison LE, Glombiewski JA, Simons LE. Enhancing Exposure Treatment for Youths With Chronic Pain: Co-design and Qualitative Approach. J Particip Med. 2023 Mar 9;15:e41292. doi: 10.2196/41292. PMID 36892929
- [Derived] Beebe JA, Kronman C, Mahmud F, Basch M, Hogan M, Li E, Ploski C, Simons LE. Gait Variability and Relationships With Fear, Avoidance, and Pain in Adolescents With Chronic Pain. Phys Ther. 2021 Apr 4;101(4):pzab012. doi: 10.1093/ptj/pzab012. PMID 33482005